CLINICAL TRIAL: NCT01697098
Title: Dexamethasone Dosing Interval: 12 or 24 Hours Apart? A Randomized,Clinical Trial
Brief Title: Dexamethasone for Preterm Labour
Acronym: PTL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Women Health Hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dexa WHH
Record Dates: First submitted 2012-09-23; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Prematurity
Keywords: Dexamethasone; preterm labour; respiratory distress
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Dyspnea | interventions — Dexamethasone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 hours Dexamethasone (Experimental): Those patient will be given 12 hours dexamethasone after randomization
  Interventions: Drug: Dexamethasone 12
- 24 hours Dexamethasone (Experimental): Those patient will be give 24 hours dexamethasone after randomization
  Interventions: Drug: Dexamethasone 24 hours

INTERVENTIONS:
Drug: Dexamethasone 24 hours
  Other Names: glucocorticoids
  Arms: 24 hours Dexamethasone
Drug: Dexamethasone 12
  Other Names: glucocorticoids
  Arms: 12 hours Dexamethasone

SUMMARY:
The investigators sought to determine whether the incidence of neonatal respiratory distress syndrome (RDS) in preterm fetuses is similar with 12- vs 24-hour dosing interval of dexamethasone.

DETAILED DESCRIPTION:
The administration of glucocorticoids to accelerate fetal lung maturity in patients with preterm delivery plays an important role for obstetrics and neonatal care. Many studies have shown that maternal administration of glucocorticoids has a significant beneficial effect in decreasing the incidence of respiratory distress syndrome (RDS) in infants delivered at 28-34 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* All patient with threatened or established preterm labor between 28 - 34 weeks attended to our emergency unit

Exclusion Criteria:

* emergent obstetric conditions like:

  * Antepartum hemorrhage in severe attack
  * Antepartum eclampsia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
respiratory distress syndrome (RDS) | 6 month
  determine whether the incidence of neonatal respiratory distress syndrome (RDS) is similar with 12- vs 24-hour dosing interval of dexamethasone.

SECONDARY OUTCOMES:
Perinatal mortality | 6 month
  Determine whether the incidence of perinatal mortality is similar with 12- vs 24-hour dosing interval of dexamethasone.

OTHER OUTCOMES:
Neonatal intensive care | 6 month
  Determine whether the incidence of admission to Neonatal intensive care is similar with 12- vs 24-hour dosing interval of dexamethasone.

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt